CLINICAL TRIAL: NCT02052882
Title: An Open Label Phase II Study of Romiplostim for Chemotherapy Induced Thrombocytopenia
Brief Title: Study of Romiplostim for Chemotherapy Induced Thrombocytopenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-132
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2023-11

CONDITIONS: Isolated Chemotherapy-induced Thrombocytopenia
Keywords: Romiplostim; Thrombocytopenia; 13-132
MeSH Terms: conditions — Thrombocytopenia | interventions — romiplostim

ARMS (1):
- Romiplostim (Experimental): All patients will begin weekly romiplostim at 2 mcg/kg, subcutaneously. The romiplostim dose will be titrated on weekly CBC/platelet counts. For titration purposes, the target platelet count is 150,000-200,000/mcL. Treatment can be held up to 16 days if a patient develops an intercurrent medical illness or symptom that is unrelated to study drug therapy.
  Treatment may be held up to 20 days if the patient unavailable for non- medical reasons, such as vacation or travel.
  Interventions: Biological: romiplostim

INTERVENTIONS:
Biological: romiplostim

SUMMARY:
This study is to determine if using weekly romiplostim injections will improve the patient's platelet count more effectively than simply waiting for the platelets to improve on its own, and if romiplostim will also allow the patient to receive at least 2 further cycles of chemotherapy without thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (18 years of age or greater) with active non-hematological cancer:

A. The patients have previously received a chemotherapy regimen including one or more of the following agents:

1. Nucleoside Analogue, including gemcitabine and fluorouracil
2. Carboplatin or cisplatin
3. Anthracycline
4. Alkylating agent
5. Other chemotherapy agents with thrombocytopenia as known common toxicity.

2. Patients who have not had any cytotoxic chemotherapy within 14 days of beginning the study.

3. Thrombocytopenia:.

A. Defined as platelet count <100,000/mcL.

B. The patient will have had at least 2 CBCs with platelet counts <100,000/mcL separated by at least 4 weeks, and no platelet count ≥100,000/mcL in the prior 6 week period, despite (1) delay, or (2) modification of chemotherapeutic regimen.

C. A platelet count of >100,000/mcL, that follows within 7 days of a platelet transfusion, will not make the patient ineligible, as long as one or more subsequent platelet counts confirms thrombocytopenia (<100,000/mcL).

D. Patients have undergone bone marrow aspirate and biopsy or peripheral blood test in the prior 3 months without evidence of leukemia or myelodysplasia by fluorescent in situ-hybridization (FISH) E. Dysplastic changes, based on morphology only, will not exclude the patient if FISH panel for MDS is normal.

4.KPS ≥ 50 or ECOG performance status ≤2 .

5.Ability to provide written informed consent.

Exclusion Criteria:

1. Patients with history of hematologic malignancies, including leukemia, myeloma, myeloproliferative disease, lymphoma, or myelodysplastic diseases.
2. Patients with known bone metastases, with evidence of corticol bone damage/lytic lesions/blastic lesions on standard imaging studies (CT/MR)
3. Anemia (Hgb <8.0 gm/dl) or leukopenia (absolute neutrophil count (ANC) <1,000/mcL). Use of red cell transfusions, erythropoietin, or G-CSF, as ordered by the managing oncology service, is acceptable and does not preclude participation.
4. Patients with underlying liver disease, such as cirrhosis or chronic hepatitis, and do not have primary or metastatic cancer in the liver will be excluded if ALT/AST >3X ULN or Total Bili >3X ULN. In the presence of primary or metastatic liver cancer, patients will be excluded if ALT/AST >5X ULN or Total Bili >5X ULN
5. Patients with a history of a prior symptomatic venous thrombotic event such, as DVT or pulmonary embolism and symptomatic arterial thrombotic events such as myocardial infarction, ischemic cerebral vascular accident or transient ischemic attack will be ineligible if they have not tolerated anticoagulation therapy. If patients remain on anticoagulation, or have completed the prescribed course of anticoagulation, they will be eligible for enrollment. A venous thrombotic event associated with a central venous catheter will not make the patient ineligible.
6. Serious concomitant medical condition that could interfere with the conduct of the clinical trial, such as unstable angina, renal failure requiring hemodialysis, or active infection requiring IV antibiotics
7. Pregnant women/lactating mothers
8. Patients unwilling to use contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01-30 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cy Wilkins, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Soff GA, Miao Y, Bendheim G, Batista J, Mones JV, Parameswaran R, Wilkins CR, Devlin SM, Abou-Alfa GK, Cercek A, Kemeny NE, Sarasohn DM, Mantha S. Romiplostim Treatment of Chemotherapy-Induced Thrombocytopenia. J Clin Oncol. 2019 Nov 1;37(31):2892-2898. doi: 10.1200/JCO.18.01931. Epub 2019 Sep 23. PMID 31545663
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Romiplostim: All patients will begin weekly romiplostim at 2 mcg/kg, subcutaneously. The romiplostim dose will be titrated on weekly CBC/platelet counts. For titration purposes, the target platelet count is 150,000-200,000/mcL. Treatment can be held up to 16 days if a patient develops an intercurrent medical illness or symptom that is unrelated to study drug therapy.
  Treatment may be held up to 20 days if the patient unavailable for non- medical reasons, such as vacation or travel.
  romiplostim
Period: Overall Study
Arm/Group | Romiplostim
Started | 60
Completed | 47
Not Completed | 13
Not completed — Not treated | 11
Not completed — Protocol Violation | 1
Not completed — Inadequate testing | 1

BASELINE CHARACTERISTICS:
Arm/Group | Romiplostim
Number analyzed (Participants) | 60
Age, Continuous [Mean (Full Range); unit: years] | 58 [27 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 46
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Platelet Counts of ≥ 100,000/mcL
Description: The primary therapeutic response is assessed by the platelet count within 3 weeks of treatment.
Time Frame: within 3 weeks after treatment
Measure: Number; unit: percentage of participants
Arm/Group | Romiplostim
Number analyzed (Participants) | 60
percentage of participants | 93

2. Secondary Outcome: Number of Participants Evaluated for Toxicity
Description: Assessment of toxicity will be based on the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Romiplostim
Number analyzed (Participants) | 60
Participants | 60

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Romiplostim
All-Cause Mortality (participants affected / at risk) | 53/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 6/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Romiplostim (N=60)
Thromboembolic event (Vascular disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Blood bilirubin increase (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT02052882/Prot_SAP_000.pdf